CLINICAL TRIAL: NCT02961270
Title: Clinical Activity of Icotinib in Patients With Advanced Non-small-cell Lung Cancer Harbouring Uncommon EGFR Mutations: a Single-arm, Prospective, Phase 2 Study
Brief Title: Icotinib in Non-small Cell Lung Cancer Patients With Uncommon EGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shengyu Zhou, Director, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMS-ZH-001
Record Dates: First submitted 2016-11-06; First posted 2016-11-10 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- icotinib (Experimental): patients will be administered study drug (icotinib) until disease progression or unacceptable toxicity
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Icotinib will be given orally 250 mg thrice per day until disease progression, or untolerated toxicity

SUMMARY:
This study aims to evaluate the efficacy of icotinib, a first generation EGFR TKI, in non-small cell lung cancer patients harboring uncommon EGFR mutation

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IIIB/IV non-small cell lung cancer
* Patients with uncommon epidermal growth factor receptor (EGFR) mutation
* Targeted-therapy-naive patients
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Evaluable target lesions according to RECIST 1.1 for tumour response assessment

Exclusion Criteria:

* Wild-type EGFR
* Positive 19 del and/or 21 L858R mutation
* Previous treatment with EGFR TKIs such as gefitinib, erlotinib, and afatinib
* Patients who have documented history of interstitial lung disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 10 months

SECONDARY OUTCOMES:
tumor response rate | 2 months
overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shengyu Zhou, MD, Study Chair — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing Key Laboratory of Clinical Study on Anticancer Molecular Targeted Drugs
Locations (1):
- Department of Medical Oncology, Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College; Beijing Key Laboratory of Clinical Study on Anticancer Molecular Targeted Drugs, Beijing, China